CLINICAL TRIAL: NCT06400316
Title: Preventing Muscle Wasting During Rheumatoid Arthritis Flares: A Randomised Controlled Trial
Brief Title: Muscle Wasting and Rheumatoid Arthritis Flares
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds Beckett University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 335887
Record Dates: First submitted 2024-01-04; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis; Muscle Atrophy
Keywords: Rheumatoid Arthritis; Muscle Atrophy
MeSH Terms: conditions — Arthritis, Rheumatoid; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: One control group will receive standard care following diagnosis of a flare of rheumatoid arthritis. The parallel group will receive a 4-week intervention involving two daily amino acid supplements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): This 'control' group will receive standard care following a flare of rheumatoid arthritis.
- Nutritional Supplementation (Experimental): This 'intervention' group will receive a 4-week intervention involving twice daily consumption of amino acid supplements.
  Interventions: Dietary Supplement: Amino Acid Supplement

INTERVENTIONS:
Dietary Supplement: Amino Acid Supplement — The intervention lasts 4-week following the rheumatoid arthritis flare. It requires twice daily consumption of amino acid supplements alongside the breakfast and lunch time meals.
  Other Names: Amino Acid Gel
  Arms: Nutritional Supplementation

SUMMARY:
People living with Rheumatoid Arthritis (RA) often present with low muscle mass compared to their healthy counterparts. This affects their mobility, overall health and quality of life. Even though low muscle mass in RA has been recognised for decades, it is still highly prevalent and very little is known about its development, progression, and potential management.

The researchers hypothesise that flares of disease activity trigger acute events of muscle wasting due to high inflammation and reduced mobility. This is commonly observed in bed rest studies and people hospitalised for various reasons. If this holds true for RA, it would point towards a stepwise development of RC and potentially allow for time-targeted management of it.

A potential method to manage it is through the use of nutritional supplements. Specifically, amino acid supplementation (commonly used by athletes or people wanting to increase muscle mass) during and shortly after a flare may counteract some of the muscle wasting and allow for better long-term mobility and quality of life for people living with RA.

This study aims to investigate aspects of muscle health changes following a disease flare-up in people with Rheumatoid Arthritis (RA) and test potential interventions to minimise any such changes. The investigators will randomly assign participants to a standard care or a nutritional supplementation group and assess aspects of body composition, muscle health, disease activity and inflammation on five occasions over a 3-month period.

DETAILED DESCRIPTION:
This study aims to investigate aspects of muscle health changes following a disease flare-up in people with Rheumatoid Arthritis (RA) and test potential interventions to minimise any such changes.

RA is the most common inflammatory arthritis manifesting mainly as joint swelling and pain, limiting mobility, and eventually leading to loss of functional capacity. RA also has severe extra-articular manifestations [1], affecting several tissues in the body including skeletal muscle [2]. People living with RA often present with an adverse body composition profile compared to the general population, characterised by low muscle mass at the presence of unchanged or even increased overall weight [3]. This condition, termed Rheumatoid Cachexia, may affect up to 2 out of 3 people with RA and associates with active disease, further reductions in mobility, and low quality of life [4].

While rheumatoid cachexia has been studied extensively, the course of its development, as well as potential causes or contributors to it are poorly understood. Inflammation, [5] as well as lifestyle factors, such as energy intake and physical activity, may contribute to the observed body composition changes [6].

People living with RA often experience flares of disease activity, where high levels of inflammation, cause an acute exaggeration of symptoms, leading to very low levels of mobility. This is commonly treated with corticosteroid injections which will rapidly reduce inflammation and allow the patient to regain mobility. However, that short period of high inflammatory load and low mobility may acutely affect muscle characteristics. Indeed, critically ill patients may lose up to 2% of skeletal muscle per day during the first week of hospitalisation [7]. This rapid decline in muscle health has been recently termed Acute sarcopenia (AS) by the European working group in sarcopenia and older persons (EWGSOP) [8]. Furthermore, recent work within this research team is currently under review (Aldrich et al., 2023 under review) demonstrating the rapid decline of muscle mass and quality in people suffering with various diseases. Additionally, corticosteroids themselves may further contribute to muscle wasting in RA [9]. Yet, the acute effects of flares and their treatment on muscle health in people with RA are not known.

Acute deterioration of muscle health following a flare may point towards a stepwise development of rheumatoid cachexia, i.e., bouts of acute deterioration that accumulate over time in steps rather than a continuous slow loss - which is the current understanding for the development of sarcopenia, the age-related muscle wasting. This would allow for target and potentially short-term interventions that could limit or even reverse muscle deterioration during a flare and help people with RA better maintain their functionality.

Exercise, and particularly resistance exercise, is the most effective way to increase muscle mass, strength, and quality. However, people during and shortly after a flare may not be willing to engage in such an intervention. Additional complexities around gym or home-based delivery, familiarisation, and safe execution render this a complex intervention with potentially limited applicability.

Nutritional supplementation on the other hand, is readily available, relatively cheap, and easy to administer. Specifically, for muscle health, amino acid supplementation, and particularly with leucine, has been shown to improve muscle mass and muscle function in older men and women [10]. Moreover, previous research has shown that these amino acid supplements do not suppress appetite, are well tolerated and easy to consume. Finally, recent unpublished data from this laboratory suggest that amino acid concentrations in the blood following consumption alongside a meal remain elevated vs placebo for over 2 hours. This indicates that consuming two supplements per day would provide sufficient amino acids to induce beneficial effects on muscle health.

Therefore, the aims of this investigation are:

1. To understand the effects of acute RA flares on muscle health
2. To assess the efficacy of amino acid supplementation vs. standard care in maintaining muscle health

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a flare of rheumatoid arthritis

Exclusion Criteria:

* Consultation with RA physician greater than 7 days before
* Allergic to supplement ingredients
* Other health conditions that affect muscle wasting; such as cancer and fibromyalgia
* Previous joint replacement surgery within the last 6 months
* Anyone with underlying kidney conditions
* Currently partaking in other research projects involving treatments, exercise or nutritional interventions for rheumatoid arthritis
* Patients who may be pregnant
* Patients who are unable to provide their own informed consent
* Patients who are unable to speak or understand English
* Participants who have a diagnosis of dementia or Alzheimer's disease
* Disabled participants who require wheelchair access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-13 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lean Tissue Mass | Scans will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Whole-body composition will be assessed by dual energy x-ray absorptiometry scans and this will provide a value for lean tissue (muscle mass) in kilograms.

SECONDARY OUTCOMES:
Quadriceps Lean Tissue Mass | Scans will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Quadriceps lean tissue mass will be assessed by dual energy x-ray absorptiometry scans focussed in the quadriceps region. Lean tissue mass in this region will be provided in kilograms.
Rectus Femoris Cross-sectional Area | Scans will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Rectus femoris will be assessed by ultrasound scans. The muscle belly will be imaged and cross-sectional area will be calculated from this image (cm2).
Handgrip Strength | Strength tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Upper-body muscle strength will be assessed by handgrip dynamometry and the value will be recorded in kilograms.
Knee Extensor Strength | Strength tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Lower-body muscle strength will be assessed on a seated knee extension resistance machine and the highest value achieved will be recorded in kilograms.
Short Physical Performance Battery | Muscle function tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Muscle function will be assessed by the Short Physical Performance Battery. This battery includes measures of gait speed, lower-limb strength/functionality and balance. The score of all tests is combined to provide a total score where a higher score indicates better muscle function.
Timed Up and Go | Muscle function tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Muscle function will be assessed by the Timed Up and Go Test. This test assesses mobility and balance. The time taken to complete standing, walking 3-metres, then returning to sit down is recorded and a shorter time indicates better functionality.
6-minute Walk Test | Muscle function tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Muscle function will be assessed by the 6-Minute Walk Test. This test assesses endurance and aerobic capacity. The total distance walked in 6 minutes is recorded and a higher score indicates greater aerobic capacity.
Plasma Amino Acid Content | Blood tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Blood plasma amino acid content (μmol/L) will be assessed at all time points using liquid chromatography mass spectrometry.
Serum Steroid Hormone Content | Blood tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Blood serum steroid hormone content (ng/ml) will be assessed at all time-points using liquid chromatography mass spectrometry.
Serum Vitamin D Content | Blood tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Blood serum vitamin D content (ng/ml)will be assessed at all time-points using liquid chromatography mass spectrometry.
Diet Recall | 24-hour diet recall tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Participants will be asked to recall their dietary intake over the preceding 24 hours to determine calorie intake.
Physical Activity | 24-hour diet recall tests will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Physical activity habits will be assessed using the International Physical Activity Questionnaire (IPAQ) (short version). Time spent sitting, walking and exercising at various intensities will be recorded in days and hours.
Physical Ability, Social Support and Interaction, Pain, Health & Mood (Quality of Life - Rheumatoid Arthritis-Specific) | Quality of life assessments will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Quality of life will be assessed using the established Rheumatoid Arthritis quality of life (RAQoL) questionnaire. This will be assessed from a series of questions which will require answers ranked from 1 (very poor) to excellent (10).
Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Interaction & Pain (Quality of Life - PROMIS-29) | Quality of life assessments will take place at baseline and 1-week, 2-weeks, 4-weeks and 12-weeks after baseline.
  Quality of life will be assessed using the Patient Reported Outcome Measures Information System (PROMIS-29) questionnaire. This will assess physical function, anxiety, depression, fatigue, sleep disturbance, ability to take part in social roles and activities, pain interference and pain intensity. All answers will be on a scale from 1 to 5 except for pain intensity which is recorded on a scale from 1 to 10. Lower scores indicate negative answers except for questions regarding physical function and pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Theocharis Ispoglou, PhD, Study Chair — Leeds Beckett University; Oliver Wilson, PhD, Study Chair — Leeds Beckett University

IPD SHARING:
Plan to Share IPD: No
Participant data will be anonymised and kept within the current research group. Participant data will not be shared with other researchers.

REFERENCES:
- [Background] Bonfiglioli KR, de Medeiros Ribeiro AC, Carnieletto AP, Pereira I, Domiciano DS, da Silva HC, Pugliesi A, Pereira LR, Guimaraes MFR, Giorgi RDN, Reis APMG, Brenol CV, Louzada-Junior P, da Cunha Sauma MFL, Radominski SC, da Mota LMH, da Rocha Castelar-Pinheiro G. Extra-articular manifestations of rheumatoid arthritis remain a major challenge: data from a large, multi-centric cohort. Adv Rheumatol. 2023 Jul 26;63(1):34. doi: 10.1186/s42358-023-00318-y. PMID 37496102
- [Background] Farrow M, Biglands J, Tanner S, Hensor EMA, Buch MH, Emery P, Tan AL. Muscle deterioration due to rheumatoid arthritis: assessment by quantitative MRI and strength testing. Rheumatology (Oxford). 2021 Mar 2;60(3):1216-1225. doi: 10.1093/rheumatology/keaa364. PMID 32910153
- [Background] Stavropoulos-Kalinoglou A, Metsios GS, Koutedakis Y, Nevill AM, Douglas KM, Jamurtas A, van Zanten JJ, Labib M, Kitas GD. Redefining overweight and obesity in rheumatoid arthritis patients. Ann Rheum Dis. 2007 Oct;66(10):1316-21. doi: 10.1136/ard.2006.060319. Epub 2007 Feb 8. PMID 17289757
- [Background] Efthymiou E, Grammatikopoulou MG, Gkiouras K, Efthymiou G, Zafiriou E, Goulis DG, Sakkas LI, Bogdanos DP. Time to Deal with Rheumatoid Cachexia: Prevalence, Diagnostic Criteria, Treatment Effects and Evidence for Management. Mediterr J Rheumatol. 2022 Sep 30;33(3):271-290. doi: 10.31138/mjr.33.3.271. eCollection 2022 Sep. PMID 36531417
- [Background] Ollewagen T, Powrie YSL, Myburgh KH, Smith C. Unresolved intramuscular inflammation, not diminished skeletal muscle regenerative capacity, is at the root of rheumatoid cachexia: insights from a rat CIA model. Physiol Rep. 2021 Nov;9(22):e15119. doi: 10.14814/phy2.15119. PMID 34806343
- [Background] Masuko K. Rheumatoid cachexia revisited: a metabolic co-morbidity in rheumatoid arthritis. Front Nutr. 2014 Nov 24;1:20. doi: 10.3389/fnut.2014.00020. eCollection 2014. PMID 25988122
- [Background] Fazzini B, Markl T, Costas C, Blobner M, Schaller SJ, Prowle J, Puthucheary Z, Wackerhage H. The rate and assessment of muscle wasting during critical illness: a systematic review and meta-analysis. Crit Care. 2023 Jan 3;27(1):2. doi: 10.1186/s13054-022-04253-0. PMID 36597123
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Lemmey AB, Wilkinson TJ, Perkins CM, Nixon LA, Sheikh F, Jones JG, Ahmad YA, O'brien TD. Muscle loss following a single high-dose intramuscular injection of corticosteroids to treat disease flare in patients with rheumatoid arthritis. Eur J Rheumatol. 2018 Sep;5(3):160-164. doi: 10.5152/eurjrheum.2018.17148. Epub 2018 Apr 2. PMID 30071930
- [Background] Ispoglou T, White H, Preston T, McElhone S, McKenna J, Hind K. Double-blind, placebo-controlled pilot trial of L-Leucine-enriched amino-acid mixtures on body composition and physical performance in men and women aged 65-75 years. Eur J Clin Nutr. 2016 Feb;70(2):182-8. doi: 10.1038/ejcn.2015.91. Epub 2015 Jun 17. PMID 26081485

DOCUMENTS (2):
  • Study Protocol (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT06400316/Prot_000.pdf
  • Informed Consent Form (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT06400316/ICF_001.pdf